CLINICAL TRIAL: NCT02040090
Title: A Prospective, Randomized, Double-Blind, Non Inferiority, Phase II/III Study of the Safety and Efficacy of Simulated Post-Exposure Prophylaxis With Kamada Human Rabies Immune Globulin (KamRAB) and Active Rabies Vaccine in Healthy Subjects
Brief Title: Phase II/III Study of the Safety and Effectiveness of HRIG With Active Rabies Vaccine in Healthy Subjects
Acronym: KAMRAB-003
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kamada, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: KAMRAB-003
Record Dates: First submitted 2013-11-28; First posted 2014-01-20 (Estimated); Results first posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2016-04

CONDITIONS: Rabies
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- KamRAB (Experimental): KamRAB 20 IU/kg body weight via IM injection, once on Day 0
  Interventions: Drug: Active rabies vaccine (US-FDA approved)
- FDA approved HRIG product (Active Comparator): Comparator product: Intramuscular (IM) injection once on Day 0 in the same manner and at the same dosage as KamRAB.
  Interventions: Drug: Active rabies vaccine (US-FDA approved)

INTERVENTIONS:
Drug: Active rabies vaccine (US-FDA approved) — A 1.0 ml dose of active vaccine (2.5 IU/ml), will be given on 5 occasions, on Days 0, 3, 7, 14, and 28 On day 0, the day when the HRIG is given, the first vaccine dose could be given within few minutes from the time of HRIG injection was given and never be administered into the same anatomical site as the HRIG.
  Other Names: RabAvert®

SUMMARY:
The purpose of this study is to: 1. Evaluate the safety and tolerability of KamRAB in comparison with Human rabies immune globulin (HRIG) comparator product. 2. To assess whether KamRAB interferes with the development of self active antibodies when given simultaneously with active rabies vaccine, as compared to the HRIG comparator product, also given in conjunction with the active rabies vaccine.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, and single period non-inferiority and safety study conducted at a single study site. Subjects were randomized into the following two groups:

Group A: KamRAB (20 IU/kg by weight [bw]) intramuscular (IM), rabies vaccine (1.0 mL; ≥2.5 IU/mL) IM Group B: Human rabies immune globulin (HRIG) Comparator product (20 IU/kg bw) IM, rabies vaccine (1.0 mL; ≥2.5 IU/mL) IM The primary endpoint was a dichotomous (0-1) variable, defined by reaching an anti-rabies immunoglobulin G (IgG) concentration ≥0.5 IU/mL on Day 14. The primary hypothesis was that the proportion of KamRAB + vaccine recipients with anti-rabies concentration ≥0.5 IU/mL on Day 14 would not be less than the corresponding proportion of HRIG Comparator subjects by as much as 0.1.

The safety and tolerability of the study treatments was assessed based on: vital signs and physical examination findings, electrocardiogram (ECG), laboratory findings (hematology, clinical chemistry, and urinalysis) and the occurrence of adverse events (AEs) after drug administration

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign an informed consent.
* Healthy male or female subjects of 18 - 75 years of age inclusive who have not previously been immunized against rabies.
* Ability to comply with completion of a home diary.
* No previous exposure to Rabies epidemic, Rabies vaccine and/or Rabies Immune globulin.
* No significant abnormalities in serum hematology, serum chemistry and serum immunogenic markers (C3, C4 and C50) according to the Principal Investigator's judgment.
* No significant abnormalities in urinalysis according to the Principal Investigator's judgment.
* No significant abnormalities in ECG per investigator judgment.
* Non-pregnant, non-lactating female subjects, whose screening pregnancy test is negative and who are using contraceptive methods deemed reliable by the investigator, or who are more than 5 years post-menopausal or surgically sterilized.
* Male subjects must be using at least one effective contraceptive method before study start and throughout the entire duration of the study.

Exclusion Criteria:

* History or laboratory evidence of immunoglobulin A deficiency.
* A history of previous administration of rabies vaccine or HRIG.
* History of live virus vaccine administration, e.g., measles vaccine, within the last 3 months.
* History of anaphylactic or anaphylactoid hypersensitivity reactions to chicken egg; history of mild allergic reactions to chicken egg, e.g., skin rash only, is not an exclusion criterion
* History of hypersensitivity reaction to any of the following components of active rabies vaccine (US-FDA approved) e.g.: neomycin, bovine gelatin, trace amounts of chicken protein, chlortetracycline, and amphotericin B and in accordance with the product insert of the vaccine.
* History of hypersensitivity reaction to any of the components in an equivalent active Rabies vaccine.
* History of allergy to blood or blood products.
* History of bleeding disorders.
* Fever at the time of the start of the infusion. (Oral temperature >38ºC.)
* Clinically significant intercurrent illnesses including: cardiac, hepatic, renal, endocrine, neurological, hematological, neoplastic, immunological, skeletal or other) that in the opinion of the investigator, could interfere with the safety, compliance or other aspects of this study.
* Evidence of active systemic infection that required treatment with antibiotics within 2 weeks of the time of drug administration.
* Evidence of uncontrolled hypertension (systolic blood pressure of >150 mm Hg, and/or diastolic blood pressure of >100 mm Hg).
* Heart rate >120/min.
* Weight > 93.75 kg
* Pregnancy and/or lactation.
* Woman of child-bearing potential not taking adequate contraception deemed reliable by the investigator.
* All types of malignancies except for basal and squamous cell (scaly or plate-like) skin cancer or situ cervical carcinoma must be in remission for a minimum of 5 years., For non-melanoma skin cancers and carcinoma in-situ of the cervix may be enrolled if treated and cured at the time of screening.
* Previous organ transplant recipient.
* Evidence of ongoing infection with Hepatitis A, C, or B, or HIV 1/2.
* Presence of psychiatric disorder, other mental disorder or any other medical disorder which might impair the subject's ability to give informed consent or to comply with the requirements of the study protocol.
* Previous enrolment in this study.
* Participation in another clinical trial within 30 days prior to baseline visit.
* Evidence of alcohol abuse or history of alcohol abuse or illegal and/or legally prescribed drugs in the past 10 years.
* History of life threatening allergy, anaphylactic reaction, or systemic response to human plasma derived products.
* Known hypersensitivity to any of the ingredients or excipients of the study drugs.
* Any other factor that, in the opinion of the investigator, would prevent the subject from complying with the requirements of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Matson, M.D., Principal Investigator — Prism Research Inc
Locations (1):
- Prism Research Inc, Saint Paul, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- KamRAB: KamRAB 20 IU/kg body weight via IM injection, once on Day 0
  Active rabies vaccine (US-FDA approved): A 1.0 ml dose of active vaccine (2.5 IU/ml), will be given on 5 occasions, on Days 0, 3, 7, 14, and 28
- FDA Approved Commercially Available HRIG Product: Comparator product: IM injection once on Day 0 in the same manner and at the same dosage as KamRAB.
  Active rabies vaccine (US-FDA approved): A 1.0 ml dose of active vaccine (2.5 IU/ml), will be given on 5 occasions, on Days 0, 3, 7, 14, and 28
Period: Overall Study
Arm/Group | KamRAB | FDA Approved Commercially Available HRIG Product
Started | 59 | 59
Completed | 56 | 57
Not Completed | 3 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- HRIG Comparator Product: FDA Approved Commercially Available HRIG Product: IM injection once on Day 0 in the same manner and at the same dosage as KamRAB.
  Active rabies vaccine (US-FDA approved): A 1.0 ml dose of active vaccine (2.5 IU/ml), will be given on 5 occasions, on Days 0, 3, 7, 14, and 28
- Total: Total of all reporting groups
Arm/Group | KamRAB | HRIG Comparator Product | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (16.15) | 46.3 (14.5) | 44.8 (15.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 22 | 21 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 57 | 53 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Difference Between KamRAB and HRIG Comparator, in the Proportions of Subjects With Serum Anti-rabies IgG Antibody Concentration ≥ 0.5 IU/mL
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | KamRAB | HRIG Comparator Product
Number analyzed (Participants) | 56 | 58
Participants | 55 | 58
Statistical Analysis 1: Comparison: KamRAB vs HRIG Comparator Product; The null hypothesis was that Cp ≤ -0.1; Test type: Non-Inferiority or Equivalence — We will reject the null hypothesis at the one-sided 5% significance level, and conclude that Cp > -0.1, if the lower bound of an exact 90% binomial confidence interval (CI) exceeds0.1. A sample size of 53 in each group provides 80% power to reject the null hypothesis; Mean Difference (Net) = -0.018, 90% CI 2-sided [-0.082 to 0.031]

ADVERSE EVENTS:
Time Frame: From signature of informed consent (ICF) to 185 days (post 8 half lives of product)
Arm/Group | KamRAB | FDA Approved Commercially Available HRIG Product
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 1/59 | 0/59
Other Adverse Events (participants affected / at risk) | 48/59 | 51/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KamRAB (N=59) | FDA Approved Commercially Available HRIG Product (N=59)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Intraductal proliferative breast lesion that was "moderate" in intensity, considered "not related" to study drug by the Principal Investigator, and was ongoing at the end of the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KamRAB (N=59) | FDA Approved Commercially Available HRIG Product (N=59)
Headache (Nervous system disorders) | 8 (8) | 9 (10)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 8 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (6)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (3)
Dizziness (Nervous system disorders) | 3 (3) | 2 (3)
Presyncope (Nervous system disorders) | 4 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 2 (3) | 2 (3)
Injection site pain (General disorders) | 29 (59) | 43 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
agreement disclosure that restricts the right of the PI to discuss or publish trial results after the trial is completed